CLINICAL TRIAL: NCT05991674
Title: A Prospective Study to Investigate Contact Sensitization Using Classic and Machine Learning Techniques
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Andreas Syggros Hospital of Venereal and Dermatological Diseases (Other)
Responsible Party: Principal Investigator, GEORGIA KOKLA, Chief Administrative Secretary, Andreas Syggros Hospital of Venereal and Dermatological Diseases
Other Study IDs: 131/2023
Record Dates: First submitted 2023-07-27; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Allergic Contact Dermatitis
Keywords: Contact Sensitization; Patch Test; Machine Learning
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — Patch Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allergic Contact Dermatitis Patients
  Interventions: Diagnostic Test: patch test for diagnosing allergic contact dermatitis

INTERVENTIONS:
Diagnostic Test: patch test for diagnosing allergic contact dermatitis — European Baseline Series (EBS) System of allergens

SUMMARY:
The goal of this study is to look into the patterns of sensitization to figure out how allergic contact dermatitis (ACD), individual susceptibility, and patient characteristics are connected. The joint application of classic statistics and machine learning methods will reveal the relationship between contact dermatitis expressions and several clinical characteristics.

ELIGIBILITY:
Inclusion Criteria:

-

Eligible patients were adults diagnosed with dermatitis who had a positive patch test result on the chemical panel of Baseline Series of Allergens.

Exclusion Criteria:

-

Although there is no consensus for the definitive exclusion criteria from a patch testing, most studies agree that the chronic use of anti-inflammatory treatments, corticosteroids, and cyclosporine, high UV exposure and other chronic dermatoses are factors that might produce false- positive or false- negative results and thus should be avoided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patch test findings from 80 ACD patients will be gathered at the National Reference Center for Occupational Dermatoses "Andreas Syggros" Hospital's Laboratory for Patch Testing.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
MOAHLFAP index | Clinical examination at baseline (0h)
  The MOAHLFAP index included characteristics of patients such as M (male), O (occupational dermatitis (OD)), A (atopic dermatitis (AD)), H (hand dermatitis (HD)), L (leg dermatitis (LD)), F (face dermatitis (FD)), A (age 40+), and P (at least one positive). Further on, we have used the criterion of trunk dermatitis (TD) and generalized dermatitis in our patients. This index contributes to the group description, stratifying the results as to the presence of sensitization prevalence and provides a multifunctional analysis in order to estimate the risk of sensitization (for example, being male with occupational contact dermatitis)
International Contact Dermatitis Research Group (ICDRG) scale | 48 hours (Day 2) and 72 hours (Day 3) after the application of patch test
  According to the International Contact Dermatitis Research Group (ICDRG) guidelines, the skin reactions are assessed as positive/allergic in terms of intesity and morphology lesions on a scale of (i) weak +, (ii) strong ++, and (iii) extreme +++, while everything else as negative (including also the irritant reactions).This is assessed as the patch test result.
Antera 3D camera (Miravex, Dublin, Ireland) | 0h (baseline), 48 hours (Day 2) and 72 hours (Day 3) after the application of patch test
  The skin condition is evaluated by the Antera 3D camera (Miravex, Dublin, Ireland) at baseline (0h), 48h and 72h after the first exposure to allergens. Antera 3D uses an innovative optical method and complex mathematical algorithms to acquire images in three dimensions. This makes it possible to extract data from images related to the three-dimensional shape of the skin, which allows the monitoring of changes over time. Hemoglobin concentration, skin texture and elevation were assessed with Antera 3D software (Miravex, Dublin, Ireland). The indications were recorded in arbitrary units.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgia Gogkla, Athens, Attica, Greece